CLINICAL TRIAL: NCT03644680
Title: Changes in Adaptive Immune Responses and Effector Cell Responses Upon Nasal Allergen Exposure - a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Ass.Prof.Dr.med. Josef Toth, Associate Professor, Doctor of Medicine, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: MUViennaIK18
Record Dates: First submitted 2018-07-26; First posted 2018-08-23 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2018-11

CONDITIONS: Allergic Rhinitis; Allergic Inflammation
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: In this single-center, randomized, placebo-controlled, double-blind study a total of 36 patients will be recruited into this study on a voluntary basis and will be randomised to receive a nasal challenge with either birch pollen extract or placebo.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nasal Provocation with Birch Extract (Experimental): Birch allergic patient receiving 3 consecutive nasal challenges with birch extract (Allergopharma). Total dose of 1.5ug of Bet v 1 per challenge
  Interventions: Diagnostic Test: Nasal Provocation with Birch Extract
- Nasal Provocation with NaCl 0.9% (Placebo Comparator): Birch allergic patient receiving 3 consecutive nasal challenges with sterile NaCl 0.9%. Total dose of 100ul per nostril per challenge
  Interventions: Other: Nasal Provocation with NaCl 0.9%

INTERVENTIONS:
Diagnostic Test: Nasal Provocation with Birch Extract — Nasal spray containing birch extract from Allergopharma
  Arms: Nasal Provocation with Birch Extract
Other: Nasal Provocation with NaCl 0.9% — Nasal spray containing sterile sodium chloride 0.9%
  Arms: Nasal Provocation with NaCl 0.9%

SUMMARY:
IgE-associated allergy is a hypersensitivity disease affecting more than 25% of the population in industrialised countries. The recognition of allergen by immunoglobulin E (IgE) plays a central role in the cause of allergic diseases. Both seasonal and nasal provocation studies have demonstrated the rise in specific IgE after allergen exposure. Additionally changes in other clinical and immunological parameters (e.g. nasal blockage, mast cell and basophil sensitivity, various cytokines or T cell profiles) in response to allergen exposure have been described. However the time sensitive interplay of these various factors such as the relationship between rise in IgE levels and change in basophils sensitivity or cytokine profiles is not yet fully understood. Clarifying how these various factors interact and contribute to immunological responses to allergen, is crucial for the development of new therapeutic approaches.

The investigators aim to address these questions through a study following 36 Birch allergic patients after provocation with allergen or placebo over a peroid of 6 weeks to 1 year.

DETAILED DESCRIPTION:
Rational of the Study

Previous studies on the dynamics of the in vivo clinical and immunological responses to nasal allergen have focused on particular parameters but have not addressed the kinetics of the interplay between the different factors (i.e. allergen-specific IgE levels, local IgE and mediator production, basophil sensitivity, cutaneous sensitivity). The investigators therefore propose a randomized double-blind placebo controlled study where The investigators challenge patients intranasally with allergen extract and then closely monitor both clinical and immunological immune responses over a period of 4 months. After this a further 4 visits will take place before and after the birch season.

The investigators will look at immediate and late phase immune responses to birch pollen extract nasal challenge outside the pollen season. Study participants will initially undergo 3 consecutive days of nasal allergen challenge and then be closely followed up for a period of 1 year. To assess clinical response to allergen exposure, The investigators will make use of the skin prick test (SPT), total nasal symptom score (TNSS), nasal endoscopy and Peak Inspiratory Nasal Flow Meter (PNIF). To assess immunological responses samples including blood, nasal mucosal sampling and nasal secretions will be taken.

Study Design

In this single-center, randomized, placebo-controlled, double-blind study a total of 36 (6 for a pre study) patients will be recruited into this study on a voluntary basis and will be randomised to receive a nasal challenge with either birch pollen extract or placebo. Randomisation will be stratified according to Bet v 1 specific IgE levels to allow for equal distribution in both groups. 30 Study participants will receive nasal provocation outside of the birch pollen season with either birch pollen extract or placebo on three consecutive days and will thereafter be followed up at a regular basis for up to four months.

Initially, prior to the study in 30 patients, 6 birch pollen allergic subjects will undergo a short protocol in order to ensure that

1. The allergen concentration used for nasal provocation is sufficient to elicit a rise of IgE antibodies
2. That the titrations of the skin prick test is adequate
3. That the timing of taking nasal secretions for determination of mediators is adequate.

   Should the results from these 6 patients reveal that either nasal allergen concentration, skin test titrations or timing of nasal secretions is not adequate, an amendment will be submitted to the ethical committee.

   The shortened protocol will include 5 visits:
   * complete screening visit
   * complete visit N1
   * visit N2 without blood sampling and without nasal sampling
   * visit N3 without blood sampling and without nasal sampling
   * complete visit N7

   Screening Visit

   Procedure
   * Signing of the Informed Consent Form (Version 2.1. for initial study with short protocol, Version 1.8 (updated for extension) for main study)
   * Allocation of screening number
   * Demographic Data
   * History of allergy
   * Assessment of In- and Exclusion Criteria
   * Pregnancy test for females if requiring SPT
   * Medical history
   * Concomitant medication
   * Anterior rhinoscopy
   * Standard SPT with commercial extract from: hazel, ash, grass mix, ragweed, mugwort, D. pteronyssinus, D. farina, cat and dog dander, alternaria, cladosporium, histamine and negative control
   * Titrated skin prick test with commercial birch pollen extract
   * Blood sampling (max 60ml of heparinized blood and serum) - A part of the blood sample will be directly sent to the laboratory for analysis of basophil activation, total IgE, and specific IgE to relevant allergens. From the rest of the blood, RNA will be prepared and stored at -80°C and serum will be separated and stored at -20°C
   * nasal sampling (nasal lavage, mucosal curette sampling and nasal secretion sampling)

   Visit N0

   Requirements regarding timing: Visit N0 is scheduled between 2 weeks and 4 days before visit N1. This is only for patients that were screened more than 3 weeks before visit N1

   Procedure:
   * Blood sampling
   * Nasal specimen collection (lavage, mucosal curette sampling and nasal secretion sampling)
   * Titrated SPT
   * PNIF
   * Pregnancy test for females if the last test was more than one month ago

   Visit N1

   Procedure:
   * Reassessment of In and Exclusion Criteria (allergen-specific IgE results)
   * Randomization: Subjects will be assigned a treatment number
   * Baseline Blood sampling
   * Baseline nasal specimen collection (lavage, nasal mucosa sampling and nasal secretion sampling)
   * Baseline TNSS score
   * Adverse event (AE) recording
   * Concomitant medication
   * PNIF given to patients and explanation/demonstration of how it works. Patients will be given a paper diary to keep track of daily PNIF values (from N1 to N5). This dairy will also be used to record daily TNSS scores (N4-N5).
   * Pregnancy test
   * i.n. administration of birch pollen extract or placebo
   * Documentation of symptoms immediately after provocation
   * Blood, PNIF, nasal sampling (nasal lavage, mucosal curette sampling and nasal secretion sampling) and TNSS score, 20min, 40min, 1hr, 2hr, 4hr, 20-24hr after birch pollen extract administration (20-24 hrs time point will be performed at visit N2).
   * Nasal sampling, PNIF and TNSS score at 10min, 3hr, 5hr, 6hr, 7hr, 8hr after birch pollen extract administration
   * Titrated SPT
   * administration of rescue medication if necessary (azelastine nasal spray, desloratadin 5mg)

   Visit N2

   Requirements regarding timing:

   Visit N2 is scheduled the day after visit N1

   Procedure:
   * Blood, PNIF, nasal sampling (lavage, mucosal curette sampling and nasal secretion sampling) and TNSS score (20-24 hour time point after birch pollen extract administration in N1).
   * AE recording
   * Concomitant medication
   * i.n. administration of birch pollen extract or placebo followed by an observation period of 2 hours
   * Documentation of symptoms immediately after provocation
   * administration of rescue medication if necessary (azelastine nasal spray, desloratadin 5mg)
   * Note: in the initial 6 study subjects nasal and blood sampling will not be performed

   Visit N3

   Requirements regarding timing:

   Visit N3 is scheduled the day after visit N2

   Procedure:
   * Blood sampling before provocation
   * Nasal specimen collection before provocation (lavage, mucosal curette sampling and nasal secretion sampling)
   * TNSS score before provocation
   * Titrated SPT
   * Adverse event (AE) recording
   * Concomitant medication
   * i.n. administration of birch pollen extract or placebo
   * Documentation of symptoms immediately after provocation
   * Blood, PNIF, nasal sampling (lavage, mucosal curette sampling and nasal secretion sampling) and TNSS score 20min, 40min, 1hr, 2hr, 4hr, 20-24hr and after birch pollen extract administration (20-24 hrs time point will be performed at visit N4).
   * Nasal sampling, PNIF and TNSS score at 10min, 3hr, 5hr, 6hr, 7hr, 8hr after birch pollen extract administration
   * Administration of rescue medication if necessary (azelastine nasal spray, desloratadin 5mg)
   * Note: in the initial 6 study subjects nasal and blood sampling will not be performed

   Visit N4

   Requirements regarding timing:

   Visit N4 is scheduled the day after visit N3

   Procedure:

   • Blood, PNIF, nasal sampling (lavage, mucosal curette sampling and nasal secretion sampling) and TNSS score at 20-24hrs after administration of birch pollen extract.

   Visit N5

   Visit N5 is scheduled 14 ±4 days after visit N4:

   Procedure:
   * Blood and nasal sampling (lavage, mucosal curette and nasal secretion sampling)
   * PNIF
   * Titrated SPT
   * TNSS score
   * AE recording
   * Pregnancy test for females if the last test was more than one month ago
   * Collection of paper diary from Visit N1 to N5

   Visit N6

   Requirements regarding timing:

   Visit N6 is scheduled 14 ±4 days after visit N5

   Procedure:
   * Blood and nasal sampling (lavage, mucosal curette and nasal secretion sampling)
   * PNIF
   * Titrated SPT
   * AE recording
   * Pregnancy test for females if the last test was more than one month ago

   Visit N7

   Requirements regarding timing:

   Visit N7 is scheduled 14 ±4 days after visit N6

   Procedure:
   * Blood and nasal sampling (lavage, mucosal curette and nasal secretion sampling)
   * PNIF
   * Titrated SPT
   * AE recording
   * Pregnancy test for females if the last test was more than one month ago

   Visit N8

   Requirements regarding timing:

   Visit N8 is scheduled 14 ±4 days after visit N7

   Procedure:
   * Blood and nasal sampling (lavage, mucosal curette and nasal secretion sampling)
   * PNIF
   * Titrated SPT
   * score
   * AE recording
   * Pregnancy test for females if the last test was more than one month ago

   Visit N9

   Requirements regarding timing:

   Visit N9 is scheduled 14 ±4 days after visit N8

   Procedure:
   * Blood and nasal sampling (lavage, mucosal curette and nasal secretion sampling)
   * PNIF
   * Titrated SPT
   * AE recording
   * Pregnancy test for females if the last test was more than one month ago

   Visit N10

   Requirements regarding timing:

   Visit N9 is scheduled 14 ±4 days after visit N9

   Procedure:
   * Blood and nasal sampling (lavage, mucosal curette and nasal secretion sampling)
   * PNIF
   * Titrated SPT
   * AE recording
   * Pregnancy test for females if the last test was more than one month ago

   Visit N11 - Final Visit of Nasal Provocation Component

   Requirements regarding timing:

   Visit N11 is scheduled 28 ±4 days after visit N10

   Procedure:
   * Blood for immunological parameters and nasal sampling (lavage, mucosal curette and nasal secretion sampling)
   * PNIF
   * Titrated SPT
   * AE recording
   * Pregnancy test for females if the last test was more than one month ago

   Visit S1 (Extension - Approved by MUW Ethics Committee on the 11th of Febuary 2019)

   Requirements regarding timing: Visit S1 is scheduled 4 weeks before the predicted start of the birch season (+/- 7 days)

   Procedure:
   * Paper pollen and PNIF diary explained to patients and asked to fill in daily during the birch season
   * Blood and nasal sampling (lavage, mucosal curette and nasal secretion sampling)
   * Titrated SPT
   * AE recording
   * Pregnancy test for females if the last test was more than one month ago

   Visit S2

   Requirements regarding timing: Visit S2 is scheduled 4 weeks after the end of the birch season (+/- 7 days)

   Procedure:
   * Blood and nasal sampling (lavage, mucosal curette and nasal secretion sampling)
   * Collection paper diary
   * Observed PNIF
   * Titrated SPT
   * TNSS score at visit
   * AE recording
   * Pregnancy test for females if the last test was more than one month ago

   Visit S3

   Requirements regarding timing:

   Visit S3 is scheduled 4 weeks after visit S2 - (+/- 7 days)

   Procedure:
   * Blood and nasal sampling (lavage, mucosal curette and nasal secretion sampling)
   * Observed PNIF
   * Titrated SPT
   * TNSS score at visit
   * AE recording
   * Pregnancy test for females if the last test was more than one month ago

   Visit S4 and End of Study

   Requirements regarding timing:

   Visit S4 is scheduled 1 year after the start of the whole study (1 year after visit N0) +/- 7 days

   Procedure:
   * Blood and nasal sampling (lavage, mucosal curette and nasal secretion sampling)
   * Observed PNIF
   * Titrated SPT
   * TNSS score at visit
   * AE recording
   * Pregnancy test for females if the last test was more than one month ago
   * End of study

   Descriptions of Study procedures

   Medical history of patients, demographic data, concomitant medication Patients will be asked for their medical history including demographic data and concomitant medication, their allergic symptoms including intensity and duration and their allergic medication history.

   History of allergy and TNSS score

   Patients will be asked for occurrence of sneezing, rhinorrhoea, nasal pruritus, nasal congestion and sleep quality and to grade each symptom at each visit and keep a record at home. They will use the following symptom score method: 0 = absent; 1 = mild - present but easily tolerated; 2 = moderate - present, symptom is bothersome but not interfering with daily life activities; 3 = severe - symptom is difficult to tolerate and is interfering with daily life activities (24). In addition to this there will be a visual analogue scale of total disease burden on the form.

   Anterior rhinoscopy

   Anterior rhinoscopy will be performed once during the screening visit to exclude anatomical variances (e.g. septal deviation) or pathological changes (e.g. nasal polyps). It will be performed by using a speculum with the patient seated with the head slightly back.

   Peak Inspiratory Nasal Flow Meter (PNIF)

   The portability and ease of the PNIF provides a unique opportunity to obtain objective measurements while the patients are at home. It has also recently been validated as a study tool during nasal allergen challenge.

   Procedure:

   At visit 1 patients will be trained how to use the PNIF device (In-check, Inspiratory ﬂow meter) and will receive one to take home with them until N5. The PNIF uses a variable diameter tube calibrated directly in litres per minute along with a low inertia indicator ring. The position of the ring after an inspiratory manoeuvre indicates the maximum flow achieved. The device works when a patient inhales through the mouth or nose, this causes air to be drawn through the meter and a cursor moves along the scale to indicate the speed of inhalation. The flow rate achieved can be noted by checking the position of the cursor against the calibrated scale.

   PNIF in study conduct:

   The PNIF will be given to study participants to take home so they can keep a daily or weekly dairy (depending on the phase of the study) of their nasal airflow. They will also be asked to bring them to all study visits so observed PNIF measurements can be taken.

   Skin prick test

   4.5.1 Procedure: Allergens are inserted into the dermis of the forearm by gently pricking the skin through a drop (20ul) of an allergen-containing solution with a sterile lancet with at least 2 cm between each individual application point. 0.9% sodium chloride solution will be used as negative and histamine as positive control. In previously sensitized individuals, itchy swelling and a reddening of the skin (wheal and flare reaction) will occur within 15 minutes upon challenge with the respective allergen. After 20 minutes, allergen solutions will be wiped off and margins of the wheals will be traced with a ball point pen. Transparent tape will be bonded on the skin in order to transfer the outline of the wheal to the tape for the records. The surface of the wheals will be calculated by digital planimetry. For inclusion, wheals of at least 3 mm in diameter will be regarded as positive reactions.

   Test solutions:

   Commercially available birch pollen extract and a panel of tree and grass pollen, weed and perennial allergens (Allergopharma, Vienna, Austria) will be used at the screening visit and will be stored according to the manufacturer's instructions. As controls, sterile 0.9% NaCl solution (negative control) and histamine (positive control, Allergopharma, Vienna, Austria) will be used. They will be stored according to the manufacturer's instructions.

   SPT in study conduct:

   Screening Visit:

   A standard skin prick test with commercial birch pollen extract and a panel of tree and grass pollen, weed and perennial allergens (all Allergopharma, Vienna, Austria) as used in routine diagnostic in the allergy clinic of the ENT department will be performed to assess the patient's sensitization profile at the screening visit.

   Screening and Visits N0, N5 - N11, S1-S4 A titrated skin prick test to birch extract will be performed with increasing dilutions (dilutions will be increased by a factor of 3 up to 1:60 000 (=11 dilution steps) to determine the lowest concentration that elicits a skin response. Skin tests to all dilutions will be done in quadruplicates. Commercial positive control solution (histamine) and negative control will be done in duplicates.

   Safety precautions As a safety precaution, patients will be monitored for 30 minutes after testing. All investigations will be done in the Outpatient Clinic of the ENT-Department, where full emergency equipment is available.

   Blood sampling and measuring of immunological parameters

   Blood samples will be taken at the screening visit and at all study visits by puncture of the antecubital vein before skin testing. A maximum of 60ml per visit will be taken either heparinized (e.g. for basophil sensitivity assays) or for the preparation of serum (e.g. for assessment of total and allergen specific immunoglobulin levels or RBL assay). Serum vials will be processed and serum will be stored at -20°C. Allergen-specific IgE of blood samples of the screening visit will be measured by CAP-FEIA to assess the allergen-specific RAST-class of the patients. Measurement of total, free, and allergen-specific serum IgE, IgG, IgA and IgM will be performed either by CAP-FEIA, by microarray measurement or ELISA. The measurement will be performed at the end of the study in all collected serum samples to minimize interassay variation. Measurement of basophil responses to allergen, fMLP and anti-IgE will be performed at each visit. Briefly, basophils will be exposed to various concentrations of anti-IgE, fMLP or recombinant allergens for 15 minutes and then examined for expression of CD 63 and CD203c by means of flow cytometry. Alternatively, histamine release will be determined by commercially available histamine release kits.

   Pregnancy testing

   In female patients, pregnancy will be excluded with a standard urine pregnancy test. The test will be performed before the first skin prick test at the screening visit and afterwards once a month.

   Nasal specimen collection

   Nasal specimen collection will be performed at all visits. For every visit specimens will be collected using nasosorption FXi/PU (containing a synthetic absorptive matrix (SAM)), or a 10 cm-long plastic curette (Both devices from Hunt Developments, UK)

   Nasosorption using FXi/PU (Hunt Developments, UK):

   Under visualization, the device will be inserted into the nasal cavity and be placed along the lateral wall against the inferior turbinate. The index finger of the patient will be used to press onto the external aspects of the alar and lateral nasal cartilages to hold the device in place. After 1 minute, the devices will be removed and the fluid will be extracted by centrifugation. Supernatant will be frozen at -70°C until further analysis for the presence of allergen-specific and total Ig levels, mediator and cytokine levels.

   Mucosal mRNA sampling A 10cm nasal curette will be used. Under direct visualisation the curette will be brought to lie against the mid-inferior portion of the inferior turbinate. The curette will be pressed against the mucosal surface moved outwards 2-3 times. This motion will be repeated 2-3 times to ensure good sample collection. This curette and technique have been shown to cause no significant discomfort to patients and thus it has the advantage of no requirement for local anaesthetic. After collection Cells will be lysed in Qiagen RLT buffer and stored at -70C for later mRNA analysis.

   4.9 Intranasal challenge

   Birch pollen extract (Allergopharma, Vienna, Austria) will be freshly diluted in sterile 0.9% sodium chloride solution and will be administered using a metered pump. The allergen will be administered using a metered pump delivering 15 μl per puff to both nostrils at visit N1, N2, N3. If the patient is suffering from nasal or eye symptoms after the challenge, azelastine nasal spray or desloratadin 5mg will be supplied.

   Randomization Procedure

   At visit N1 of the main study, patients will be randomized to one of the two groups (Birch pollen extract or Placebo). Study subjects will be randomized (ratio 2:1 for provocation versus control) using the online randomization programme "randomizer" (www.meduniwien.ac.at/randomizer), which is maintained at the Institute for Medical Informatics, Statistics and Documentation at Medical University of Graz, Graz, Austria. The 2:1 ratio is chosen because the variance of Ig measurements and derived quantities is expected to be larger in the provocation group due to expected larger overall Ig levels, also see the sample size consderations later in this document.

   The randomization will be carried out by a person who is not involved in the study and has no contact with the patients to ensure that the study will be double blinded.

   Investigational products and study medication

   Birch Pollen Extract:

   Birch pollen extract (Allergopharma, Vienna, Austria) will be used for intranasal challenge. Birch pollen extract will arrive lyophilised and will be dissolved in sterile 0.9% sodium chloride. The content of Bet v 1 in the extract will be determined by immunoblotting using antibody probes specific for Bet v 1. Finally the extract will be diluted so that the final concentration of Bet v 1 will be 50 μg/ml as this concentration has previously been shown to elicit changes in specific IgE levels upon nasal challenge.

   Control solutions:

   Control solutions will comprise sodium chloride 0.9% as negative control for skin prick test and as placebo for intranasal challenge. Histamine (Allergopharma, Vienna, Austria) will be used as a positive control for the skin prick test. They will be stored according to the manufacturer's instructions.

   Concomitant medication

   General:

   All additional medication being taken by the subjects on entry to the study or at any time during the study are regarded as concomitant medication and will be documented in the Source Data File. Concomitant medications should be kept to a minimum during the study, but if considered necessary may be given if not interfering with the study protocol.

   Rescue medication:

   Although anaphylactic events are very unlikely in this study they always have to be considered possible. Therefore a complete emergency kit will be available immediately in case of anaphylactic reactions at SPT or nasal challenge. Furthermore if the patient is suffering from nasal and eye symptoms after the intranasal challenge azelastine nasal spray and/or desloratadin 5mg will be provided to ameliorate the symptoms.

   Prohibited concomitant medication:

   Subjects must remain off medications interfering with study procedures for the duration of the study. The following concomitant treatments are not permitted during this study:
   * Systemic or topical corticosteroids
   * Other immunosuppressant drugs
   * Antihistamines or disodium cromoglycate 3 days prior to visits
   * Systemic or intranasal adrenergic drugs
   * Psychopharmacological drugs
   * ACE-inhibitors or beta-blockers

   Adverse events

   An adverse event is any event during a clinical study, including intercurrent illness or accident, which impairs the well-being of the subject; it may also take the form of an abnormal laboratory value. The term adverse event does not imply a causal relationship with the study treatment.

   All subjects experiencing adverse events - whether considered associated with the use of the study treatment or not - will be monitored until symptoms subside and any abnormal laboratory value has returned to baseline, or until there is a satisfactory explanation for the changes observed, or until death, in which case a full pathology report from a qualified pathologist will be provided. All findings must be reported on an "adverse event" page in the case record form.

   All adverse events will be reported on and documented as described below. Adverse events are divided into the categories "serious" and "non-serious". This determines the procedure which must be used to report/document the adverse event.

   Definition of serious and non-serious adverse events

   A serious adverse event is:
   * Any event that is fatal or life-threatening
   * Any event that is permanently disabling
   * Any event that requires or prolongs hospitalization
   * Any event that involves cancer, congenital abnormality, or occurs as a result of overdose (application of more than the stipulated dose).

   Adverse events which do not fall into these categories are defined as non-serious.

   Assessment of severity of AE

   Regardless of the classification of an adverse event as serious or non-serious (see above), its severity must be assessed as mild, moderate or severe, according to medical criteria alone:

   Mild = does not interfere with routine activities, acceptable Moderate = interferes with routine activities Severe = impossible to perform routine activities, considered as unacceptable by the physician, requires treatment, requires discontinuation of study, or has residual effect.

   It should be noted that a severe adverse event need not be serious in nature. Regardless of severity, all serious adverse events must be reported on as below.

   Reporting/documentation of adverse events

   Adverse events are collected by spontaneous reporting.

   Reporting/documentation of serious adverse events

   All serious adverse events which occur during this study whether considered to be associated with the study medication or not, must be documented on an "Adverse event" page in the case record form.

   A follow-up report including all new information obtained on the serious event must be prepared and will be collected.

   The investigator will submit on request copies of all these reports to the ethics committee. Where necessary, investigators will inform the authorities.

   Reporting/documentation of non-serious adverse events

   These are to be documented on an "Adverse event" page in the case record form.

   Statistical analysis

   As this is a pilot study, the performed analysis are considered as explorative and hypothesis generating.

   Patient characteristics and outcome variables will be described by calculating maximum, minimum, median, mean and standard deviation for metric variables and absolute and relative frequencies for categorical variables.

   To analyse time-trajectories of IgE levels and other outcome variables, descriptive statistics as well as 95% confidence intervals for the mean will be calculated for each time-point and each treatment group separately. To account for heterogeneous baseline levels between patients, the observed outcomes for each patient will be standardized by the respective baseline values for these analyses. Further, mean differences between groups and according 95% confidence intervals will be calculated for each time-point. For graphical illustration, the individual trajectories of each patient will be plotted.

   The data observed in the skin prick test consists of a series of allergen doses and the resulting area measurements. Based on preliminary data from eight patients in previous study, an exponential model of the type Area = A*(1-exp(-λ Dose) was found to appropriately describe the dose-response relationship observed in the skin prick test. The model will be fit for of each time point in each group using a non-linear least squares algorithm. From these models, the response rate λ, the plateau area A and the 50% effective dose will be reported together with 95% confidence intervals.

   If there are missing values, all analysis will be done on an available case basis.

   Sample size considerations:

   Given the exploratory nature of the study, the sample size considerations are based on the precision of parameter estimates. The primary objective is the analysis of IgE levels across time. Date from a previous study show a relative increase of anti-Bet v 1 IgE four weeks after nasal provocation with Bet v 1 by a mean factor of 1.4 and a standard deviation of approximately 0.5 between patients. With a control antigen, the mean factor was 1.04 with a standard deviation of approximately 0.25. The maximal statistical precision for a comparison of mean values between the two groups is achieved if the allocation ratio is proportional to the ratio of standard deviations, which is 2:1 based on the previous data. Under the above assumptions on effect sizes and standard deviations, a total sample size of 30 (20:10) will provide 95% confidence intervals with a half-width of approximately 0.2 in either group. The expected half-width of a 95% confidence interval for the mean difference between groups is 0.28. (A corresponding two-sample t-test would have a power of 80% to detect a mean difference of 0.4 at a 5% significance level). For the analysis of the skin prick test, the preliminary data suggest that with a sample size of 20, the half-width of 95% confidence intervals for the 50% effective dose will be approximately 0.25 times the 50% effective dose, which is considered as sufficient precision for this pilot study. Please see appendix for graphical representation

   Ethical and legal aspects

   The study will be carried out in keeping with local legal requirements and GCP. It will be performed in accordance with the guidelines of the Declaration of Helsinki (1964), including current revisions.

   Informed consent of subject

   Before being admitted to the study, the subject must have consented to participate after the nature, scope and possible consequences of the clinical study have been explained in a form understandable to him/her. The subject must give consent in writing. The signature of the investigator will confirm the subject's consent. The patient may withdraw the consent, even without giving comments, at any time and without negative consequences for his future medical care.

   Acknowledgement/approval of the study

   Before the start of the study, the study protocol will be submitted to the Ethics committee of the medical university Vienna and the general hospital of Vienna (Borschkegasse 8b/E 06, 1090 Vienna, Austria).

   Insurance

   All subjects participating in this study will be insured at the Zürich Insurance company (Zürich-Versicherungs-Aktiengesellschaft, Schwarzenbergplatz 15, 1010 Vienna, Tel. +43 50 1255 1255; insurance number: 07229622-2).

   Confidentiality

   All subjects' names will be kept secret in the investigators files. Subjects will be identified throughout documentation and evaluation by the number allotted to them during the study. The subjects will be told that all study findings will be stored and handled in strictest confidence.

   Documentation and use of study findings

   Documentation of study findings

   All results collected during the study will be collected in a source data file and will later be transferred to the case report forms (CRFs). All entries on the case record forms will be made legibly in black or blue ink. If corrections are made to entries in the case record form, the words or figures will be ringed and a single stroke drawn through them. The correct value will be entered beside the old entry and date and the correction will be initialled. Incorrect entries must not be covered with correcting fluid or obliterated or made illegible in any way. The completed CRFs will be signed by the investigator. CRFs will be completed immediately after the final examination. The medical records upon which the CRF is based will be kept for at least 15 years.

   Use of the study findings

   The findings of this study will be published by the investigators in a scientific journal and presented in scientific meetings. The manuscript will be circulated to all co-investigators before submission.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18 to 60 years of age
* Birch pollen sensitized subjects
* Moderate to severe allergic rhinitis to birch pollen for at least two seasons according to medical history
* Sensitization to Bet v 1 (3.5 kU/L Bet v 1 specific IgE or higher as determined by UniCAP-FEIA)
* CD203c or CD63 upregulation or histamine release upon challenge with Bet v 1 in basophil activation tests (at least 20% increase in upregulated CD63 or CD203c expression or histamine release on basophils upon stimulation compared to unstimulated controls measured by flow cytometry)
* Willingness to comply with the study protocol and written informed consent
* Subjects must have a standard health care insurance
* Subjects must be available during the study period to complete all treatments and assessments

Exclusion Criteria:

* History of anaphylaxis
* Any severe chronic, malignant or general disease
* Treatment with systemic or topical (intranasal, inhaled, external) corticosteroids within the previous 2 months before the start of the study
* Treatment with antihistamines 3 days prior to the screening visit of the study
* Treatment with other immunosuppressant drugs within the previous 6 months prior to the start of the study
* Arterial hypertension or use of anti-hypertensive therapy, including beta-blockers
* Contra-indications to skin prick testing such as: skin inflammation in the test area, urticaria facticia
* Sensitisation to an allergen which is relevant during the birch pollen season (e.g., ash tree pollen, house dust mite etc)
* Pregnant, lactating or sexually active women with childbearing potential who are not using a medically accepted birth control method
* A mental condition rendering the subject unable to understand the nature, scope and possible consequences of the study, and/or evidence of an uncooperative attitude
* Participation in another clinical trial within one month prior to the study; however participation during the previous month solely in the form of blood donation and/or without other interventions will be accepted
* Known alcohol or drug addiction or abuse
* Risk of non-compliance with the study procedure
* Active asthma currently necessitating treatment
* Previous immunotherapy with birch pollen
* Nasal polyps, history of chronic sinusitis or substantial deviation of the nasal septum

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2019-10-04 (Actual); Study Completion 2019-10-04 (Actual)

PRIMARY OUTCOMES:
Allergen Specific IgE Rise | 1 Year
  To assess changes of allergen specific IgE levels after challenge with Birch pollen extract

SECONDARY OUTCOMES:
IgE Levels in Nasal Secretions | 1 Year
  To assess changes in allergen-specific IgE levels in nasal secretions after nasal provocation with birch pollen extract
Total IgE Levels | 1 Year
  To assess changes in total IgE levels after nasal provocation with birch pollen extract
Assessing Immunoglobin Isotypes | 1 Year
  To assess changes in allergen-specific and total IgA, IgD, IgG (including subtypes) and IgM levels in sera and nasal secretions after nasal provocation with birch pollen extract by ELISA
Changes in TH2 Cytokine patterns. | 1 Year
  To assess changes in TH2 cytokine patterns in sera and nasal secretions after nasal provocation with birch pollen extract. This we be determined by ELISA or Luminex assay which will mean cytokine measurements will have the same units of measure.
IgE Production | 1 Year
  To assess presence and changes in IgE production (i.e., by RT-PCR with primers specific for IgE) in nasal mucosa
Subjective Symptom Assessment | 1 Year
  To assess changes in nasal symptoms using the validated scoring system, Total Nasal Symptom Score (TNSS). On this scale 4 nasal symptoms are assessed namely sneezing, rhinorrhea, nasal itching and nasal blockage on a scale of 0 (no symptoms) 1 (mild symptom burden), 2 (moderate symptom burden) or 3 (severe symptom burden). The scores a totaled and a score out of 12 is produced. Higher values represent greater allergic symptom burden.
Nasal Blockage | 1 Year
  To objectively assess the degree of change in nasal blockage by PNIF
Skin Response | 1 Year
  To assess the changes in skin reactivity to allergen in a titrated skin prick test to birch pollen extract

CONTACTS AND LOCATIONS:
Overall Officials: Josef Toth, MD, Principal Investigator — ENT Specialist
Locations (1):
- 8H1.02, ENT Lab, Department of Otorhinolaryngology, Vienna General Hospital, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wuthrich B, Schindler C, Leuenberger P, Ackermann-Liebrich U. Prevalence of atopy and pollinosis in the adult population of Switzerland (SAPALDIA study). Swiss Study on Air Pollution and Lung Diseases in Adults. Int Arch Allergy Immunol. 1995 Feb;106(2):149-56. doi: 10.1159/000236836. PMID 7819743
- [Background] Bischoff SC. Role of mast cells in allergic and non-allergic immune responses: comparison of human and murine data. Nat Rev Immunol. 2007 Feb;7(2):93-104. doi: 10.1038/nri2018. PMID 17259966
- [Background] Valent P, Bettelheim P. The human basophil. Crit Rev Oncol Hematol. 1990;10(4):327-52. doi: 10.1016/1040-8428(90)90009-h. No abstract available. PMID 2278641
- [Background] Galli SJ, Tsai M, Piliponsky AM. The development of allergic inflammation. Nature. 2008 Jul 24;454(7203):445-54. doi: 10.1038/nature07204. PMID 18650915
- [Background] Sadan N, Rhyne MB, Mellits ED, Goldstein EO, Levy DA, Lichtenstein LM. Immunotherapy of pollinosis in children: investigation of the immunologic basis of clinical improvement. N Engl J Med. 1969 Mar 20;280(12):623-7. doi: 10.1056/NEJM196903202801201. No abstract available. PMID 4180015
- [Background] Yunginger JW, Gleich GJ. Seasonal changes in IgE antibodies and their relationship to IgG antibodies during immunotherapy for ragweed hay fever. J Clin Invest. 1973 May;52(5):1268-75. doi: 10.1172/JCI107294. PMID 4735589
- [Background] Naclerio RM, Adkinson NF Jr, Moylan B, Baroody FM, Proud D, Kagey-Sobotka A, Lichtenstein LM, Hamilton R. Nasal provocation with allergen induces a secondary serum IgE antibody response. J Allergy Clin Immunol. 1997 Oct;100(4):505-10. doi: 10.1016/s0091-6749(97)70143-x. PMID 9338545
- [Background] Niederberger V, Ring J, Rakoski J, Jager S, Spitzauer S, Valent P, Horak F, Kundi M, Valenta R. Antigens drive memory IgE responses in human allergy via the nasal mucosa. Int Arch Allergy Immunol. 2007;142(2):133-44. doi: 10.1159/000096439. Epub 2006 Oct 19. PMID 17057411
- [Background] Eckl-Dorna J, Pree I, Reisinger J, Marth K, Chen KW, Vrtala S, Spitzauer S, Valenta R, Niederberger V. The majority of allergen-specific IgE in the blood of allergic patients does not originate from blood-derived B cells or plasma cells. Clin Exp Allergy. 2012 Sep;42(9):1347-55. doi: 10.1111/j.1365-2222.2012.04030.x. PMID 22925321
- [Background] Shi FC, Huang HS, Huang MJ, Juang JH, Chen GW. [Cushing's syndrome with pregnancy. Report of three cases]. Changgeng Yi Xue Za Zhi. 1992 Dec;15(4):226-33. Chinese. PMID 1295659
- [Background] Galli SJ, Tsai M. IgE and mast cells in allergic disease. Nat Med. 2012 May 4;18(5):693-704. doi: 10.1038/nm.2755. PMID 22561833
- [Background] Eckl-Dorna J, Froschl R, Lupinek C, Kiss R, Gattinger P, Marth K, Campana R, Mittermann I, Blatt K, Valent P, Selb R, Mayer A, Gangl K, Steiner I, Gamper J, Perkmann T, Zieglmayer P, Gevaert P, Valenta R, Niederberger V. Intranasal administration of allergen increases specific IgE whereas intranasal omalizumab does not increase serum IgE levels-A pilot study. Allergy. 2018 May;73(5):1003-1012. doi: 10.1111/all.13343. Epub 2017 Dec 12. PMID 29083477
- [Background] Campana R, Moritz K, Marth K, Neubauer A, Huber H, Henning R, Blatt K, Hoermann G, Brodie TM, Kaider A, Valent P, Sallusto F, Wohrl S, Valenta R. Frequent occurrence of T cell-mediated late reactions revealed by atopy patch testing with hypoallergenic rBet v 1 fragments. J Allergy Clin Immunol. 2016 Feb;137(2):601-609.e8. doi: 10.1016/j.jaci.2015.08.042. Epub 2015 Oct 28. PMID 26518092
- [Background] Leaker BR, Malkov VA, Mogg R, Ruddy MK, Nicholson GC, Tan AJ, Tribouley C, Chen G, De Lepeleire I, Calder NA, Chung H, Lavender P, Carayannopoulos LN, Hansel TT. The nasal mucosal late allergic reaction to grass pollen involves type 2 inflammation (IL-5 and IL-13), the inflammasome (IL-1beta), and complement. Mucosal Immunol. 2017 Mar;10(2):408-420. doi: 10.1038/mi.2016.74. Epub 2016 Sep 28. PMID 27677865
- [Background] van Hage-Hamsten M, Pauli G. Provocation testing with recombinant allergens. Methods. 2004 Mar;32(3):281-91. doi: 10.1016/j.ymeth.2003.08.007. PMID 14962763
- [Background] Egger C, Lupinek C, Ristl R, Lemell P, Horak F, Zieglmayer P, Spitzauer S, Valenta R, Niederberger V. Effects of nasal corticosteroids on boosts of systemic allergen-specific IgE production induced by nasal allergen exposure. PLoS One. 2015 Feb 23;10(2):e0114991. doi: 10.1371/journal.pone.0114991. eCollection 2015. PMID 25705889
- [Background] Kim YW, Singh A, Shannon CP, Thiele J, Steacy LM, Ellis AK, Neighbour H, Gliddon DR, Hickey PLC, Larche M, Tebbutt SJ. Investigating Immune Gene Signatures in Peripheral Blood from Subjects with Allergic Rhinitis Undergoing Nasal Allergen Challenge. J Immunol. 2017 Nov 15;199(10):3395-3405. doi: 10.4049/jimmunol.1700378. Epub 2017 Oct 18. PMID 29046347
- [Background] Shamji MH, Bellido V, Scadding GW, Layhadi JA, Cheung DK, Calderon MA, Asare A, Gao Z, Turka LA, Tchao N, Togias A, Phippard D, Durham SR. Effector cell signature in peripheral blood following nasal allergen challenge in grass pollen allergic individuals. Allergy. 2015 Feb;70(2):171-9. doi: 10.1111/all.12543. PMID 25377909
- [Background] Dhariwal J, Cameron A, Trujillo-Torralbo MB, Del Rosario A, Bakhsoliani E, Paulsen M, Jackson DJ, Edwards MR, Rana BMJ, Cousins DJ, Hansel TT, Johnston SL, Walton RP; MRC-GSK Strategic Alliance Consortium. Mucosal Type 2 Innate Lymphoid Cells Are a Key Component of the Allergic Response to Aeroallergens. Am J Respir Crit Care Med. 2017 Jun 15;195(12):1586-1596. doi: 10.1164/rccm.201609-1846OC. PMID 28085492
- [Background] Kleiner S, Braunstahl GJ, Rudrich U, Gehring M, Eiz-Vesper B, Luger TA, Steelant B, Seys SF, Kapp A, Bohm M, Hellings PW, Raap U. Regulation of melanocortin 1 receptor in allergic rhinitis in vitro and in vivo. Clin Exp Allergy. 2016 Aug;46(8):1066-74. doi: 10.1111/cea.12759. Epub 2016 Jun 15. PMID 27196703
- [Background] Eguiluz-Gracia I, Bosco A, Dollner R, Melum GR, Lexberg MH, Jones AC, Dheyauldeen SA, Holt PG, Baekkevold ES, Jahnsen FL. Rapid recruitment of CD14(+) monocytes in experimentally induced allergic rhinitis in human subjects. J Allergy Clin Immunol. 2016 Jun;137(6):1872-1881.e12. doi: 10.1016/j.jaci.2015.11.025. Epub 2016 Feb 4. PMID 26851967
- [Background] Tworek D, Kuna P, Mlynarski W, Gorski P, Pietras T, Antczak A. MIG (CXCL9), IP-10 (CXCL10) and I-TAC (CXCL11) concentrations after nasal allergen challenge in patients with allergic rhinitis. Arch Med Sci. 2013 Oct 31;9(5):849-53. doi: 10.5114/aoms.2013.37198. Epub 2013 Aug 26. PMID 24273568
- [Background] Baroody FM, Detineo M, Naclerio RM. Unilateral nasal allergic reactions increase bilateral sinus eosinophil infiltration. J Appl Physiol (1985). 2013 Nov 1;115(9):1262-7. doi: 10.1152/japplphysiol.00547.2013. Epub 2013 Aug 22. PMID 23970539
- [Background] Downie SR, Andersson M, Rimmer J, Leuppi JD, Xuan W, Akerlund A, Peat JK, Salome CM. Symptoms of persistent allergic rhinitis during a full calendar year in house dust mite-sensitive subjects. Allergy. 2004 Apr;59(4):406-14. doi: 10.1111/j.1398-9995.2003.00420.x. PMID 15005764
- [Background] Boelke G, Berger U, Bergmann KC, Bindslev-Jensen C, Bousquet J, Gildemeister J, Jutel M, Pfaar O, Sehlinger T, Zuberbier T. Peak nasal inspiratory flow as outcome for provocation studies in allergen exposure chambers: a GA2LEN study. Clin Transl Allergy. 2017 Sep 17;7:33. doi: 10.1186/s13601-017-0169-4. eCollection 2017. PMID 28932387
- [Background] Focke M, Marth K, Valenta R. Molecular composition and biological activity of commercial birch pollen allergen extracts. Eur J Clin Invest. 2009 May;39(5):429-36. doi: 10.1111/j.1365-2362.2009.02109.x. PMID 19302561